CLINICAL TRIAL: NCT00576901
Title: "An Open Label Study to Assess the Effect of Neoadjuvant Treatment With Docetaxel + Xeloda + Avastin on Pathological Response Rate in Inflammatory or Locally Advanced Breast Cancer"
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Xeloda (Capecitabine) and Docetaxel in Patients With Inflammatory or Locally Advanced Breast Cancer.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sample for statistical analysis of results could not be recruited within the specified timeframe upon retirement of the original principal investigator.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20561
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Docetaxel; Capecitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: Docetaxel; Drug: Xeloda

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 15mg/kg iv on day 1 of each 3 week cycle
Drug: Docetaxel — 75mg/m2 iv on day 1 of each 3 week cycle
Drug: Xeloda — 2000mg/m2 po on days 1-15 of each 3 week cycle

SUMMARY:
This single arm study will assess the efficacy and safety of combination first-line treatment with docetaxel + Xeloda + Avastin in patients with inflammatory or locally advanced breast cancer. Patients will receive 3-weekly cycles of Avastin (15mg/kg i.v. on day 1 of each cycle), docetaxel (75mg/m2 i.v. on day 1 of each cycle, after Avastin) and Xeloda (2000mg/m2 p.o. on days 1-15 of each cycle). Four cycles of chemotherapy are planned, plus an optional additional two cycles; after chemotherapy patients will be assessed for surgery. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >=18 years of age;
* HER2-negative, locally advanced (stage II or III) or inflammatory cancer of the breast;
* ECOG performance status 0-1.

Exclusion Criteria:

* metastatic disease (stage IV);
* previous treatment for breast cancer;
* evidence of CNS metastasis;
* current or recent (within 10 days of first dose of Avastin) use of aspirin (>325mg/day) NSAIDs or full dose anticoagulants for therapeutic purposes;
* clinically significant cardiovascular disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Madrid, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab+Docetaxel+Capecitabine: Participants received bevacizumab 15 milligrams per kilogram (mg/kg), intravenously (IV), on Day 1; docetaxel 75 mg per square meter (mg/m^2), IV, on Day 1; and capecitabine 2000 mg/m^2, orally, on Days 1-15. This cycle was repeated every 3 weeks for a total of 4 cycles. If all 4 cycles were tolerated, participants then completed an additional 2 cycles, for a maximum of 6 cycles of study treatment.
Period: Overall Study
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Started | 23
Completed | 20
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Disease course | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population. The ITT population included all enrolled participants.
Groups:
- Bevacizumab+Docetaxel+Capecitabine: Participants received bevacizumab 15 mg/kg, IV, on Day 1; docetaxel 75 mg/m^2, IV, on Day 1; and capecitabine 2000 mg/m^2, orally, on Days 1-15. This cycle was repeated every 3 weeks for a total of 4 cycles. If all 4 cycles were tolerated, participants then completed an additional 2 cycles, for a maximum of 6 cycles of study treatment.
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.96 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Pathological Complete Response (pCR)
Description: pCR was defined as the absence of viable tumor cells, as determined by standard histologic procedure, in the tumor specimen (including regional lymph nodes) obtained at surgery. In order to minimize evaluation bias, tumor specimens were analyzed by both a central and local pathologist. The number of participants with pathological tumor stage 0 (pT0) and regional lymph nodes stage 0 (pN0) at surgery was determined. pCR was defined as the number of participants with pT0 and pN0 at surgery divided by the total number of participants with pathological tumor stage data collected.
Time Frame: At time of surgery, after receiving up to 6 cycles of treatment (average of 12 to 18 weeks)
Population: Evaluable Response (ER) Population: study-eligible participants who completed at least 2 treatment cycles; had lesions evaluated using the same technique at baseline and at least once after receiving the second treatment cycle; and had no major protocol deviation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Number analyzed (Participants) | 20
percentage of participants | 0

2. Secondary Outcome: Percentage of Participants Achieving an Overall Response of Complete Response (CR) or Partial Response (PR)
Description: The percentage of participants with a best overall response of CR or PR according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must have decreased to normal (short axis less than [<]10 millimeters [mm]). No new lesions. PR was defined as greater than or equal to (≥) 30 percent (%) decrease under baseline of the sum of diameters of all target lesions. The short aixs was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Day 1 of Cycles 1-6
Population: ER population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Number analyzed (Participants) | 20
percentage of participants | 80

3. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival was defined as the time from the date of informed consent until the date disease progression was identified, or the date of death from disease progression, whichever occurred first.
Time Frame: Cycles 1-6
Population: The application of a statistical model for the analysis of disease-free survival was not feasible as the sample size required for statistical analysis could not be recruited within the time established in the protocol and the study was terminated.
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of informed consent until the date of death due to any cause.
Time Frame: Cycles 1-6
Population: The application of a statistical model for the analysis of disease-free survival is not feasible as the sample size required for statistical analysis could not be recruited within the time established in the protocol and the study was terminated.
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Number analyzed (Participants) | 0

5. Secondary Outcome: Percentage of Participants Undergoing Breast-Conserving Surgery
Description: The percentage of participants who were able to undergo breast-conserving surgical procedures (segmentectomy plus lymphadenectomy or quadrantectomy plus lymphadenectomy) rather than non-breast conserving procedures (radical mastectomy or modified-radical mastectomy) following 4 or more treatment cycles.
Time Frame: Following Cycle 6
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Number analyzed (Participants) | 23
percentage of participants | 26.09

ADVERSE EVENTS:
Time Frame: Throughout study
Description: The safety population included all participants who received at least 1 dose of study treatment.
Arm/Group | Bevacizumab+Docetaxel+Capecitabine
Serious Adverse Events (participants affected / at risk) | 2/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Docetaxel+Capecitabine (N=23)
Neutropenia (Blood and lymphatic system disorders) | 1
Disease progression (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab+Docetaxel+Capecitabine (N=23)
Alopecia (Skin and subcutaneous tissue disorders) | 9
Nausea (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 14
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 11
Vomiting (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 9
Headache (Nervous system disorders) | 3
Nail toxicity (Skin and subcutaneous tissue disorders) | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 2
Mucous membrane inflammation (General disorders) | 5
Cystitis (Infections and infestations) | 1
Upper abdominal pain (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 6
Neurotoxicity (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 2
Vaginal bleeding (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hypersensitivity (Immune system disorders) | 2
Abnormal liver function test (Investigations) | 1
Mastitis (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 1
Palpebral edema (Eye disorders) | 1
Urinary tract infections (Infections and infestations) | 1
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Laryngitis (Infections and infestations) | 1
Odynophagia (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.